CLINICAL TRIAL: NCT02885337
Title: Fit-Joints: Getting Fit for Hip or Knee Replacement, A Pilot Randomized Control Trial
Brief Title: Fit-Joints: Getting Fit for Hip or Knee Replacement
Acronym: Fit-Joints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Alexandra Papaioannou, Professor of Medicine, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1565
Record Dates: First submitted 2016-08-09; First posted 2016-08-31 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
Keywords: Frail Elderly; Arthroplasty; Frailty
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Frailty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): Patients in the control arm will receive usual care which may include the recommendation to attend fitness classes before surgery, however these patients will not receive the more intensive assessment/intervention of the physiotherapist and other intervention components. Control participants will be asked pre-operatively and post-operatively to indicate whether or not they exercise, take protein or vitamin supplements.
  For participants in intervention and control groups will, 1) we will monitor the YMCA attendance and 2) participants will be instructed on the completion a dietary intake log (including days of the week and weekend days) that indicate the type of food and amount over a four-day period in order to calculate energy and micronutrient consumption.
  Interventions: Other: Usual Care
- Multi-Modal Frailty Intervention (Experimental): Exercise: A physiotherapist will develop an individualized exercise program and schedule appointments with patients at a physiotherapist clinic. Participants will be offered free YMCA membership.
  Cognitive-behavioural Change Strategy(CBCS) and education: Throughout the intervention, CBCS and education about exercise, hip or knee arthroplasty and osteoarthritis will be administered.
  Protein Supplement: Participants will be provided with 1-2 daily supplements (containing 20-40 gram protein, 1.5 g β-Hydroxy β-Methylbutyrate /serving) to be taken with a meal or on activity days within 3-hours of exercise.
  Vitamin D: All participants in the intervention arm will be provided with a supply of Vitamin D3 (1000 IU/day tablets) for the duration of the intervention period.
  Medication Review: A geriatrician will review the medications for patients in the intervention arm.
  Interventions: Other: Multi-Modal Frailty Intervention; Other: Usual Care

INTERVENTIONS:
Other: Multi-Modal Frailty Intervention — Exercise: A physiotherapist will develop an individualized exercise program and schedule appointments with the patient at a physiotherapist clinic. Participants will be offered free YMCA membership.
  Cognitive-behavioural Change Strategy(CBCS) and education: Throughout the intervention, CBCS and education about exercise, hip or knee arthroplasty and osteoarthritis will be administered.
  Protein Supplement: Participants will be provided with 1-2 daily supplements (containing 20-40 gram protein, 1.5 g β-Hydroxy β-Methylbutyrate /serving) to be taken with a meal or on activity days within 3-hours of exercise.
  Vitamin D: All participants in the intervention arm will be provided with a supply of Vitamin D3 (1000 IU/day tablets) for the duration of the intervention period.
  Medication Review: A geriatrician will review the medications for patients in the intervention arm.
  Arms: Multi-Modal Frailty Intervention
Other: Usual Care — Patients in the control arm will receive usual care which may include the recommendation to attend fitness classes before surgery, however these patients will not receive the more intensive assessment/intervention of the physiotherapist and other intervention components. Control participants will be asked pre-operatively and post-operatively to indicate whether or not they exercise, take protein or vitamin supplements.
  For participants in intervention and control groups will, 1) we will monitor the YMCA attendance and 2) participants will be instructed on the completion a dietary intake log (including days of the week and weekend days) that indicate the type of food and amount over a four-day period in order to calculate energy and micronutrient consumption.

SUMMARY:
Osteoarthritis leads to reduced independence and quality of life. Total hip replacement is a successful and cost-effective surgical intervention to relieve pain and improve functioning in patients with osteoarthritis. Research has shown that preoperative health status strongly predicts outcomes including physical function and hospitalization length after hip replacement surgery. Frail patients, in particular, are at greater risk of poor postoperative outcomes and could potentially benefit from interventions targeting an improvement in their health status prior to undergoing a hip or knee replacement surgery. Partnering with the YMCA and a multi-disciplinary team of healthcare providers, this pilot trial will examine the feasibility of a multi-modal intervention for frail patients that includes a supervised exercise program, vitamin D and protein supplementation, and a medication review. The results of this feasibility study will guide the design of a future multi-centre study, which if successful, could be developed into a routine model of care that is implemented in joint replacement programs across Ontario and ultimately improving the lives of frail seniors undergoing hip or knee replacement.

DETAILED DESCRIPTION:
Study Design: The proposed study is a pilot randomized controlled trial comparing a pre-operative multi-modal intervention and standard care among pre-frail/frail patients undergoing total hip or knee replacement surgery. Pre-frail (score of 1 or 2) or frail (score of 3-5; Fried Frailty Phenotype) patients, ≥ 60 years undergoing elective unilateral total hip or knee replacement after at least 3 months will be recruited from the practices of 8 orthopedic surgeons (Hamilton Arthroplasty Group).

A research assistant (RA) will conduct the eligibility screening at the Regional Joint Assessment Program (Hamilton Health Sciences) and St. Joseph's Healthcare, Hamilton, ON during an appointment (3-9 months prior to surgery). Patients with renal insufficiency, a neuromuscular disorder, active cancer or any inflammatory arthritis will be excluded.

Stratified block randomization will be used to randomly allocate participants to the intervention or usual care arms of the study. The allocation sequence will be computer generated using Statistical Analysis Software (SAS) 9.3. Once the study RA confirms the patient's eligibility, and obtain consent, the RA will inform the research coordinator (RC) who will randomize the participant using Red Cap randomization list. Then the RC will call the participants to inform them if they fall in the intervention or control group and arrange the first visit.

Multi-Modal Frailty Intervention (3-9 months). Exercise: A Registered physiotherapist will develop an individualized exercise program and schedule appointments with the patient at home including goal setting discussion. Participants will be offered free YMCA membership to participate in the IN Motion program.The IN Motion program is designed for older adults and include gentle fit, hydrotherapy and walk fit classes along with health education sessions. Participants will be taught how to monitor their own heart rate and level of exertion using the Borg Rating of Perceived Exertion 10-point Scale. All participants will be encouraged to exercise at least 3 times per week for 45-60 minutes either at home and/or at YMCA IN Motion classes. The home exercise will incorporate aerobic, resistance training, flexibility and balance components. Patients will be provided with and asked to keep an exercise log-book.

Cognitive-behavioral Change Strategy and education:

Cognitive Behavioral Change Strategies (CBCS) may be an effective way to facilitate coaching strategies to increase participant exercise levels. In the current study, modules will be presented to participants in the event that they express any barriers to exercise. These barriers will vary based on: the individual, environment, and previous exercise behaviors. Throughout the intervention, CBCS will be performed and administered by the physiotherapist prior to the participants scheduled surgery. The administration of the modules will be dependent on the challenges that the participants express in relation to exercise (i.e., lack of time, motivation, social support, etc.). A definition of each strategy will be given to the participant; the physiotherapist will then work through a worksheet with the participant.

Protein Supplement: Participants will be provided with 1-2 daily supplements (containing 20-40 gram protein, 1.5 g β-Hydroxy β-Methylbutyrate /serving) to be taken with a meal or on activity days within 3-hours of exercise.

Vitamin D: All participants in the intervention arm will be provided with a supply of Vitamin D3 (1000 IU/day tablets) for the duration of the intervention period.

Medication Review: After randomization, a geriatrician will review the medications for patients in the intervention arm and provide written recommendations to the participant's family doctor.

Control arm: Patients in the control arm will receive usual care which may include the recommendation to attend fitness classes before surgery; however these patients will not receive the more intensive assessment/intervention of the physiotherapist and other intervention components. Control participants will be asked pre-operatively and post-operatively to indicate whether or not they exercise, take protein or vitamin supplements.

For participants in intervention and control groups will, 1) be monitored for their YMCA attendance and 2) be instructed on the completion a dietary intake log that indicate the type of food and amount over a four-day period in order to calculate energy and micronutrient consumption. Then a RA will call the participants to collect their food intake.

ELIGIBILITY:
Participants will be included if they are: 1) ≥ 60 years old; 2) pre-frail (score of 1 or 2) or frail (score of 3-5; Fried Frailty Phenotype); 3) receiving elective unilateral hip or knee replacement; and 4) waiting time to surgery is estimated to be between 3 to 9 months. Participants will be excluded if reported having: 1) renal insufficiency (due to potential contraindication of additional protein); 2) neuromuscular disorder; 3) active cancer; or 4) any inflammatory arthritis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-08; Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, an average of two years
  4 patient/month
Retention Rate | Through study completion, an average of two years
  target ≥ 70%
Data Collection completion | Through study completion, an average of two years
  target ≥ 70%
Proportion of recruited patients | Through study completion, an average of two years
  target ≥ 70%
Refusal Rate | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
  target ≥ 70%

SECONDARY OUTCOMES:
GERAS Fit Frailty Index to measure frailty | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
Oxford Hip or Knee Score to measure pain and function | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
Sarc-F to measure sarcopenia | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
European Quality of Life-5 Dimensions to measure health related quality of life | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
Mini-Cog Test to measure cognitive function | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
Older Americans Resources and Services Questionnaire to measure basic and instrumental activity of daily life | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
Number of Hospital admission (or readmissions) | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
Number of visits to Healthcare providers | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
Number of medications and supplements | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
Discharge Destination | 6 weeks post-op and 6 months post-op
Number of Falls | 1 week pre-op, 6 weeks post-op, 6 months post-op
Number of Adverse Events | 1 week pre-op, 6 weeks post-op, 6 months post-op
Serum 25-Hydroxy Vitamin D | Baseline and 6 weeks post-op
Serum Pre-Albumin | Baseline and 6 weeks post-op
Short Performance Physical Battery | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
Fried Frailty Phenotype | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op
Length of stay after surgery | 6 weeks post-op, 6 months post-op
Length of stay - rehabilitation | 6 weeks post-op, 6 months post-op
Surgical Complications | 6 weeks post-op, 6 months post-op
Number of ER visits | Baseline, 1 week pre-op, 6 weeks post-op, 6 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, MD,MSc, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - McMaster University - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okpara C, Negm A, Adachi JD, Armstrong D, Atkinson S, Avram V, de Beer J, Hladysh G, Ioannidis G, Kennedy C, Hewston P, Lau A, Lee J, Richardson J, Marr S, Panju A, Petruccelli D, Thabane L, Winemaker M, Papaioannou A. Getting fit for hip and knee replacement: The Fit-Joints multimodal intervention for frail patients with osteoarthritis - a pilot randomized controlled trial. J Frailty Aging. 2025 Apr;14(2):100028. doi: 10.1016/j.tjfa.2025.100028. Epub 2025 Mar 4. PMID 40042971
- [Derived] Negm AM, Kennedy CC, Ioannidis G, Gajic-Veljanoski O, Lee J, Thabane L, Adachi JD, Marr S, Lau A, Atkinson S, Petruccelli D, DeBeer J, Winemaker M, Avram V, Deheshi B, Williams D, Armstrong D, Lumb B, Panju A, Richardson J, Papaioannou A. Getting fit for hip and knee replacement: a protocol for the Fit-Joints pilot randomized controlled trial of a multi-modal intervention in frail patients with osteoarthritis. Pilot Feasibility Stud. 2018 Jul 20;4:127. doi: 10.1186/s40814-018-0316-2. eCollection 2018. PMID 30038794